CLINICAL TRIAL: NCT02536898
Title: Norwegian Capture the Fracture Initiative
Acronym: NoFRACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Asker & Baerum Hospital (Other); Drammen sykehus (Other); Haukeland University Hospital (Other); Molde Hospital (Other); St. Olavs Hospital (Other); University Hospital of North Norway (Other); University of Oslo (Other); Norwegian University of Science and Technology (Other)
Responsible Party: Principal Investigator, Lene Bergendal Solberg, Prof. Dr. Med., Oslo University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2015/334
Record Dates: First submitted 2015-04-30; First posted 2015-09-01 (Estimated); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Hip Fracture; Vertebral Fracture; Other Low-trauma Fracture
MeSH Terms: conditions — Hip Fractures; Spinal Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fracture liaison service (Experimental): * Information, assessment & lifestyle advice
  * refer to DXA scan, except patients with dementia, difficulties laying on the back or short life exp.
  * Blood samples
  * Sufficient intake of Vitamin D & calcium, combined with physical activity will be recommended with lifestyle advice (smoking & alcohol intake)
  * Patients With Hip, Vertebral or two or more low-trauma fractures are recommended treated with anti-osteoporosis drug
  * Other fractures, treatment recommended if FRAX score≥20% for major fracture & T-score≤-1.5
  * Fracture patients with reduced kidney function will be treated with anti-RANKL
  * Anti-osteoporosis drug prescribed by hospital physician
  * Follow-up phone call after 3 months and visit to talk with coordinating nurse after 1 year
  * Patients with spine or femoral neck T-scores≤-3.5, >2 severe vertebral fractures & those who suffer a second fracture while using anti-osteoporosis drug, will be referred for further examination and teriparatide treatment will be considered
  Interventions: Other: Fracture Liaison Service
- Current treatment (Other): Treatment as offered before intervention.
  Interventions: Other: Current treatment

INTERVENTIONS:
Other: Fracture Liaison Service
  Arms: Fracture liaison service
Other: Current treatment
  Arms: Current treatment

SUMMARY:
The main aim is to assess the effectiveness of introducing a standardized intervention program for treatment of patients with a fragility fracture as measured by changes in the fracture rates and the mortality.

DETAILED DESCRIPTION:
A fracture liaison service model of care is widely recommended but data on its effectiveness regarding reduced risk of recurrent fracture and fracture related mortality are scarce. The investigators therefore aim to assess the risk of subsequent fractures and mortality after a clinical fracture in patients who present to hospitals with a standardized intervention program. Seven Norwegian hospitals will be Stepped Wedge Cluster Randomized to a standardized intervention program with startup date between May 2015 and Jan 2016. The intervention will last throughout 2018 with follow-up throughout 2019. Outcomes before and after the intervention will be compared and each hospital will act as its own control. The effect of the intervention will be measured by using national patient registries on fractures and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Low-energy fracture

Exclusion Criteria:

* finger fracture, toe fracture, face fracture, skull fracture

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94260 (Actual)
Dates: Start 2015-05; Primary Completion 2020-01 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
Fragility fracture | 4 years
  Incidence of fragility fractures per 10,000 person-years (distal forearm fractures, proximal humerus fractures and hip fractures)

SECONDARY OUTCOMES:
Mortality | 4 years
  Total number of deaths during four years after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Lars Nordsletten, PhD, Study Director — Oslo University Hospital
Locations (7):
- Norway (7):
  - Haukeland University Hospital, Bergen
  - Drammen Hospital, Drammen
  - Molde Hospital, Molde
  - Oslo University Hospital, Oslo
  - Bærum Hospital, Sandvika
  - University Hospital of North Norway, Tromsø
  - St. Olavs University Hospital, Trondheim

REFERENCES:
- [Derived] Andreasen C, Solberg LB, Basso T, Borgen TT, Dahl C, Wisloff T, Hagen G, Apalset EM, Gjertsen JE, Figved W, Hubschle LM, Stutzer JM, Elvenes J, Joakimsen RM, Syversen U, Eriksen EF, Nordsletten L, Frihagen F, Omsland TK, Bjornerem A. Effect of a Fracture Liaison Service on the Rate of Subsequent Fracture Among Patients With a Fragility Fracture in the Norwegian Capture the Fracture Initiative (NoFRACT): A Trial Protocol. JAMA Netw Open. 2018 Dec 7;1(8):e185701. doi: 10.1001/jamanetworkopen.2018.5701. PMID 30646281